CLINICAL TRIAL: NCT03773601
Title: Objective Sleep Behavior in Relation to a Nigth Competition in Athletes: a Pilot Study.
Brief Title: Objective Sleep Behavior in Relation to a Nigth Competition in Athletes.
Acronym: Sleep Profiler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sleep Profiler and athletes
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Athlete; Sleep Deprivation
Keywords: Sleep; Athlete; Sleep Profiler
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes (Experimental): Athletes will undergo a 4-days sleep monitoring with the use of the Sleep Profler. At the same time, they will fill the Total Quality of Recovery (TQR) scale and the Pittsburgh Sleep Quality Index (PSQI).
  Interventions: Other: Sleep Profiler; Other: PSQI; Other: TQR

INTERVENTIONS:
Other: Sleep Profiler — A 4-days sleep monitoring with the use of the Sleep Profiler. Data on objective sleep behavior will be collected.
Other: PSQI — Fill the Pittsburgh Sleep Quality Index (PSQI) for the subjective evaluation of sleep.
Other: TQR — Fill the Total Quality of Recovery Scale (TQR), every morning for 4 consecutive days, to collect data on subjective perception of recovery,

SUMMARY:
Sleep is a crucial factor for athletes' health and recovery. Many variables are able to negatively influence the sleep of top-level athletes, such as: anxiety, long travels, high volume or high-intensity training period, and a nigth competition too. Therefore, the aim of this pilot study is to evalute how sleep quality changes in relation to a late nigth competition in athletes.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age between 18 and 45
* sport activity for > or = to 8 hours/week.
* signed informed consent

Exclusion Criteria:

* smoking
* part-time or shift worker.
* Use of medications able to influence sleep
* any medical conditions (injury) contraindicating physical exercise as diagnosed by a sports medicine physician

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | From the 1st to the 4th nigth of monitoring
  Evaluation of the changes in Sleep Efficiency, evaluated by the Sleep Profiler, before (1st and 2nd nigths) and after (3rd and 4th nigths) a nigth competition.

SECONDARY OUTCOMES:
TQR | From the 1st to the 4th nigth of monitoring
  Evaluation of the changes in the subjective perception of recovery, evaluated with the Total Quality of Recovery Scale (TQR), before (1st and 2nd nigths) and after (3rd and 4th nigths) a nigth competition.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacopo Antonino Vitale, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided